CLINICAL TRIAL: NCT03110991
Title: A Randomized Controlled Trial on the Efficacy of a Cognitive-behavioral Intervention Via a Smartphone App for Caregivers With Depressive Symptoms
Brief Title: Cognitive-behavioral Intervention Via a Smartphone App for Depressive Symptoms in Caregivers
Acronym: App Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); Ministry of Work and Welfare - Xunta de Galicia (Other Government)
Responsible Party: Principal Investigator, Fernando Lino Vázquez González, Tenured Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PSI2016-79041-P
Record Dates: First submitted 2017-03-22; First posted 2017-04-12 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Depression
Keywords: Depression; Depressive symptoms; Prevention; Non-professional caregivers; App
MeSH Terms: conditions — Depression; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive-behavioral intervention via App (Experimental): The participants of the two experimental groups will receive a cognitive-behavioral intervention for depression prevention via a smartphone App, adapted from an indicated depression prevention program for caregivers in face-to-face group format developed by our research team, based on the model by Lewinsohn, Hoberman, Teri, & Hautzinger (1985), which has proven to be efficacious in the prevention of the onset of new major depressive episodes and the decrease of depressive symptoms both short- and long-term (Vázquez et a., 2014, 2016). In both groups the intervention administered via App will consist of 5 modules.
  Interventions: Behavioral: Multicomponent Cognitive Behavioral Intervention administered via a smartphone App (CCIA)
- Cognitive-behavioral intervention via App + multiconference (Experimental): Additionally, this experimental group will receive phone group conference calls during four 30 minute-sessions.
  Interventions: Behavioral: Multicomponent Cognitive Behavioral Intervention administered via a smartphone App+ telephone contact via conference call (CCIA+CC)
- Usual care (No Intervention): Individuals assigned to this group will receive no intervention or material, but they will have unrestricted access to any routine medical or psychological care that they might want to seek to treat depressive symptoms.The use of such treatments will be recorded.

INTERVENTIONS:
Behavioral: Multicomponent Cognitive Behavioral Intervention administered via a smartphone App (CCIA) — Multicomponent Cognitive Behavioral Intervention administered via a smartphone App (CCIA)
  Arms: Cognitive-behavioral intervention via App
Behavioral: Multicomponent Cognitive Behavioral Intervention administered via a smartphone App+ telephone contact via conference call (CCIA+CC) — Multicomponent Cognitive Behavioral Intervention administered via a smartphone App+ telephone contact via conference call (CCIA+CC)
  Arms: Cognitive-behavioral intervention via App + multiconference

SUMMARY:
Major depression is a common disorder among non-professional caregivers, and it can be disabling and costly. Although there are effective psychological interventions to prevent depression, most of them involve in-person treatment. New technologies have the potential to overcome the barriers this format presents, which limit accessibility to such interventions. The main objective of this project is to evaluate the effectiveness of a cognitive-behavioral intervention in the prevention of depression, administered through a smartphone application (App), both with and without telephone contact through multiconferencing. Secondary objectives are: (a) test the moderating or mediating effect of the variables in the theoretical model underlying the intervention; (b) analyze the variables that are predictors of intervention outcomes; (c) analyze the acceptability and satisfaction with interventions. A randomized controlled trial will be perform. Caregivers with clinically significant depressive symptoms who do not meet the diagnostic criteria for depressive episode will be included. Recruitment of 174 participants is planned, with random allocation to one of the three conditions (58 participants per intervention): (a) a cognitive-behavioral intervention administered via a smartphone App (CCIA); (b) a cognitive-behavioral intervention administered via a smartphone App + telephone contact via conference call (CCIA+CC); (c) attention control group (ACG). Both interventions will be administered in 5 modules via an App for Smartphones and one group additionally will receive telephone contact via conference call in group format during 4 sessions of 30 minutes. These phone sessions will be recorded to assess the therapists adherence to the intervention protocols. All participants will be evaluated at pre and posttreatment, and 1-, 3-, 6- and 12-month follow-up by trained interviewers who will be blind to the aims of the study, the interventions employed, and the group to which any given participant belongs. Incidence of depression will be examined as the primary measure, with secondary measures being depressive symptoms, symptoms related to the model (pleasant activities, negative thoughts and social contacts) and the acceptability of and satisfaction with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Serves as an informal caregiver for dependent family member
* Dependence is recognized by the Xunta de Galicia
* Commitment to participate in all assessments
* A CES-D score ≥ 16
* Not suffering from a depressive episode
* Provides informed consent
* Has a Smartphone

Exclusion Criteria:

* Having received psychological or pharmacological treatment in the previous two months
* To present other conditions that may act as confounders (e.g., symptoms due to substance use)
* Presenting serious psychological or medical disorders that require immediate intervention (e.g., suicidal ideation) or prevent study implementation (e.g., significant cognitive impairment)
* The dependent has a serious or terminal prognosis for the next 14 months
* Planning a change of address or institutionalization of the family member for the next 14 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Major depressive episode to post-treatment (6 weeks), and follow-ups at 1, 3, 6 and 12 months | Pre- and post-intervention (6 weeks) with follow-ups at 1, 3, 6, and 12 months
  The presence of a major depressive episode will be assessed with the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders-5, DSM-5® -Clinician Version (SCID-5-CV; First, Williams, Karg, & Spitzer, 2015). This is a semi-structured interview that provides DSM-5 diagnosis and must be administered by a specialized professional. It includes diagnostic assessment of depressive disorder, bipolar disorder, schizophrenia and other psychotic disorders, substance use disorders, anxiety disorders, obsessive-compulsive disorder, posttraumatic stress disorders, attention deficit and hyperactivity disorder, adaptative disorders, and it allows screening for 17 additional disorders. For this study the module corresponding to major depressive episode was use. The interrater reliability (Kappa) ranges from .70 y 1.00.

SECONDARY OUTCOMES:
Change from baseline depressive symptomatology to post-treatment (6 weeks), and follow-ups at 1, 3, 6 and 12 months | Pre- and post-intervention (6 weeks) with follow-ups at 1, 3, 6, and 12 months
  Depressive symptoms as measured by the Center for Epidemiological Studies Depression Scale [CES-D] (Radloff,1977; Spanish version of Vazquez, Blanco, & Lopez, 2007). This 20-item scale is self-administered and assesses depressive symptoms. The person evaluates each item based on how often they have experienced it in the last week using a Likert scale with four response options ranging from 0 (rarely or none of the time) to 3 (most of the time).The total score ranges from 0 to 60, and higher scores correspond to greater depressive symptomatology. Internal consistency (Cronbach's alpha) of the scale ranges from .85 and .90, with .89 for the Spanish version (Vazquez et al.,2007 and 2014).

OTHER OUTCOMES:
Socio-demographic characteristics | Pre-intervention
  Sociodemographic characteristics were collected via the Care Characteristics and Status of Caregiver questionnaire. This questionnaire was developed in a previous study (Vázquez et al., 2014, 2016), and assesses the sociodemographic characteristics (sex, age, marital status, social class, family monthly income per household, level of education, main occupation and area of residence), and the care situation (number of persons cared for, relationship with the persona cared for, age and sex of the person cared for, disease of the person cared for, time of care, and hours a day of care) of non professional caregivers.
Change from baseline Automatic negative thoughts to post-treatment (6 weeks) | Pre- and post-intervention (6 weeks)
  The occurrence of automatic negative thoughts will be assessed through the 30-item Automatic Negative Thoughts Questionnaire (ATQ-N, Hollon and Kendall, 1980). The subject must indicate the frequency for which a number of thoughts have suddenly arisen in their mind over the last week on a five-point scale from 1 (never) to 5 (always). Scores range between 30 and 150, and there is a direct relationship between the score and the frequencies of certain types of thoughts, with a higher score indicating more negative thoughts experienced by the subject. The internal consistency for the ATQ-N subscale is .96.
Change from baseline Pleasant activities to post-treatment (6 weeks) | Pre- and post-intervention (6 weeks)
  The pleasant activities will be assessed via the List of Pleasant Activities for Caregivers (LAA). It includes 40 activities to evaluate the pleasant activities that the caregivers have performed during the last week. It consists of a pleasant activities list, where the participants indicate whether or not a certain activity is pleasant to them, if they performed it during the last week, and the number of times it was carried out (developed and used in a previous study; Vázquez et al., 2016). In the previous study it showed an internal consistency of .89.
Change from baseline Social contacts to post-treatment (6 weeks) | Pre- and post-intervention (6 weeks)
  To evaluate the participants' weekly social contacts we will use the Register of Social Networking (developed and used in the previous study by Vazquez et al., 2016) that asks the participants to report the number of people they had daily contact with.
Number of dropouts | During the intervention sessions (5 weeks)
  We will construct a registry of the number of dropouts from each group to assess their response to the interventions over the duration of the study.
Treatment adherence | During the intervention sessions (5 weeks)
  Treatment adherence will be assessed by recording the number of meetings each caregiver attends and whether they complete homework assignments.
Satisfaction with the service received | Post-intervention (6 weeks)
  Participant satisfaction with the service received will be evaluated upon intervention completion. We will use the Client Satisfaction Questionnaire ([CSQ-8]; Larsen, Attkisson, Hargreaves, & Nguyen, 1979; Spanish version Vazquez, Torres, & Otero, 2009). It is an 8-item scale with 4 possible answers and a final ranking score ranging from 8 to 32, where a higher score implies greater satisfaction with the service received. It is a widely used tool with an internal consistency between .83 and .93 (Attkisson & Greenfield, 2004).

CONTACTS AND LOCATIONS:
Overall Officials: Fernando L. Vázquez González, Ph.D., Principal Investigator — Tenured Professor
Locations (1):
- Research Group on Mental Health and Psychopatology, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attkisson CC; Greenfield TK. The UCSF Client Satisfaction Scales: I. The Client Satisfaction Questionnaire-8. In Maruish ME, editor, The use of psychological testing for treatment planning and outcomes assessment. 3rd ed. Volume 3. Mahwah, NJ: Lawrence Erlbaum Associates; 2004. p. 799-811.
- [Background] First MB, Williams, JBW, Karg RS, Spitzer RL. Structured Clinical Interview for DSM-5 Disorders, Clinician Version (SCID-5-CV). Arlington, VA: American Psychiatric Association; 2015.
- [Background] Hollon SD; Kendall PC. Cognitive self-statements in depression: development of an Automatic Thought Questionnaire. Cognitive Ther Res 1980; 4: 383-395.
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Lewinsohn PM, Hoberman H, Teri L, Hautzinger M. An integrative theory of depression. In Reiss S, Bootzin RR, editors, Theoretical issues in behaviour therapy. New York: Academic Press; 1985, p. 313-359.
- [Background] Radloff LS. A CES-D scale: a self-report depression scale for research in thegeneral population. Appl Psychl Meas 1977; 1: 385-401.
- [Background] Vazquez FL, Blanco V, Lopez M. An adaptation of the Center for Epidemiologic Studies Depression Scale for use in non-psychiatric Spanish populations. Psychiatry Res. 2007 Jan 15;149(1-3):247-52. doi: 10.1016/j.psychres.2006.03.004. Epub 2006 Dec 1. PMID 17141880
- [Background] Vázquez FL; Hermida E; Torres A; Otero P; Blanco V; Díaz O. Eficacia de una intervención preventiva cognitivo conductual en cuidadoras con síntomas depresivos elevados. Behav Psychol 2014; 22: 77-94.
- [Background] Vazquez FL, Torres A, Blanco V, Otero P, Diaz O, Ferraces MJ. Long-term Follow-up of a Randomized Clinical Trial Assessing the Efficacy of a Brief Cognitive-Behavioral Depression Prevention Intervention for Caregivers with Elevated Depressive Symptoms. Am J Geriatr Psychiatry. 2016 Jun;24(6):421-32. doi: 10.1016/j.jagp.2016.02.050. Epub 2016 Feb 27. PMID 27067068
- [Background] Vázquez FL, Torres A, Otero P. CSQ-8 Castilian (TMS.047). Available in: http://www.CSQscales.com; 2009.
- [Derived] Vazquez FL, Torres A, Diaz O, Paramo M, Otero P, Blanco V, Lopez L. Cognitive behavioral intervention via a smartphone app for non-professional caregivers with depressive symptoms: study protocol for a randomized controlled trial. Trials. 2018 Jul 31;19(1):414. doi: 10.1186/s13063-018-2793-2. PMID 30064466